CLINICAL TRIAL: NCT03020667
Title: An Observational Cohort Study in Japan to Assess the Patterns of Product Use and Changes in Health Outcomes Associated With the Use of HeatSticks With the IQOS Tobacco Heating System
Brief Title: Japanese Post-Market Cohort Study
Status: Terminated | Type: Observational
Why Stopped: The study was terminated due to excessive attrition rates.
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: P1-PMC-01-JP
Record Dates: First submitted 2016-11-17; First posted 2017-01-13 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Smoking; Tobacco Product
Keywords: Cigarette; IQOS; Nicotine-containing product; Tobacco
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IQOS Users: The criteria defining an "IQOS user" are listed in the section "Eligibility".
- Cigarette (CC) Smokers: The criteria defining a "CC smoker" are listed in the section "Eligibility".

SUMMARY:
The objectives and endpoints of this study were analyzed in the study population of adults eligible to purchase tobacco products. The study was planned to describe the patterns of use of tobacco and nicotine containing products and self-reported health outcomes and health related events in CC (Cigarette) smokers and IQOS users in Japan.

The initial study record (posted on ClinicalTrials.gov) included a clinical sub-study designed to estimate population level differences in the biomarkers of exposure and clinical risk endpoints among IQOS users, CC smokers and never-smokers. However, due to low recruitment and retention of subjects, the clinical sub-study was terminated in May 2017, and for the same reasons the main study was terminated in March 2018. The study protocol was updated to remove the clinical sub-study objectives. The study initially included 18 outcome measures. Due to study termination leading to a shortened follow-up period and a smaller sample size, only 7 of these outcome measures could be assessed and the other outcome measures planned were either unattainable or uninformative.

DETAILED DESCRIPTION:
This was a prospective, observational, cohort study of adults, eligible to purchase tobacco products in Japan. The study described the patterns of use of tobacco and nicotine containing products in CC smokers and IQOS users.

For IQOS users, the date of initiation of IQOS use was the trigger for all study assessments in the study. However the process was different for CC smokers for whom assessment timing was based on the date of enrollment. IQOS users were enrolled into the study at least two months after initiating use of IQOS (to ensure adoption of IQOS), but less than 12 months after initiating use of IQOS. The study assessments started at the next appropriate study time point after enrollment. Participants were recruited from consumer databases and/or through advertisement. Responses from all eligible participants in the study were collected online using computer assisted self-interviews (CASIs). The questionnaires included demographic information, tobacco use questionnaire including detailed product use and intention to stop tobacco- and nicotine-containing product use, lifestyle assessments, social-economic status, risk perception, nicotine dependence, urge to smoke, as well as self-reported health outcomes. IQOS users were also administered the Modified Cigarette Evaluation Questionnaire, and Self-Reported Changes Questionnaire. The CASIs were administered at the enrollment and quarterly for the first 18 months (at Months 3, 6, 9, 12, 15 and 18).

The study initially was planned to recruit 2,000 IQOS users and 2,000 cigarette (CC) smokers in 4 annual waves (500 IQOS users and 500 CC smokers per wave) and to be followed up to a maximum of 60 months. The first wave of recruitment competed in March 2017. During wave 2 recruitment the study was terminated. A total of 599 IQOS users and 525 CC smokers were enrolled. There was 1 reported protocol deviation in IQOS users, the participant had been using IQOS for 15 months. Due to study termination, only data collected for wave 1 was analyzed.

As this study was observational by design and was conducted in a post-market setting, adverse event (AE) reporting followed the Sponsor's established post-market Safety Surveillance Procedures for spontaneously reported events. IQOS users were reminded of the product quality complaints (including AEs) hotline that is available for all IQOS consumers in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Adult tobacco users in Japan (at least 20 years of age)
* The participant is Japanese
* Participant is able to understand the information provided in the Informed Consent form (ICF)
* Signed ICF
* Willing to participate in the study and has access to the internet
* For IQOS users:

  * Is currently using IQOS with HeatSticks
  * Has used at least 100 HeatSticks with IQOS in their lifetime, and
  * Has used IQOS with HeatSticks for 2 months or more
* For CC smokers:

  * Is currently using CC
  * Is not currently using IQOS with HeatSticks, and
  * Has used at least 100 CC in their lifetime

Exclusion Criteria:

* Tobacco industry employees
* Employed by the Sponsor, CRO or Clinical Site
* For IQOS users:

  * More than 12 months of IQOS use

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (female or male) Japanese IQOS users and CC smokers.
Sampling Method: Non-Probability Sample
Enrollment: 1124 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kunihiko Uwatoko, MD, Principal Investigator — Uwatoko Clinic; Pierpaolo Magnani, Study Chair — Philip Morris Products S.A.
Locations (1):
- Uwatoko Clinic, Ōzone, Nagoya, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 525 CC smokers and 599 IQOS users were enrolled, 70 IQOS users initiated IQOS 3 months ago, 191 IQOS users initiated IQOS 6 months ago, 264 IQOS users initiated IQOS 9 months ago, 73 IQOS users initiated IQOS 12 months ago, and 1 IQOS user initiated IQOS 15 month ago.
  Note: only data collected of wave 1 participants was analyzed.
Pre-assignment Details: CC smokers: based on the date of enrollment. IQOS users: based on date of initiation of IQOS use (IQOS use time).
Groups:
- CC Smokers: The criteria defining a "CC smoker" are listed in the section "Eligibility".
- IQOS Users: 3 Months IQOS Use Time; IQOS Users: 6 Months IQOS Use Time; IQOS Users: 9 Months IQOS Use Time; IQOS Users 12 Months IQOS Use Time; IQOS Users 15 Months IQOS Use Time: The criteria defining a "IQOS user" are listed in the section "Eligibility".
Period: At Month 3
Arm/Group | CC Smokers | IQOS Users: 3 Months IQOS Use Time | IQOS Users: 6 Months IQOS Use Time | IQOS Users: 9 Months IQOS Use Time | IQOS Users 12 Months IQOS Use Time | IQOS Users 15 Months IQOS Use Time
Started | 525 | 70 | 0 | 0 | 0 | 0
Completed | 215 | 70 | 0 | 0 | 0 | 0
Not Completed | 310 | 0 | 0 | 0 | 0 | 0
Period: At Month 6
Arm/Group | CC Smokers | IQOS Users: 3 Months IQOS Use Time | IQOS Users: 6 Months IQOS Use Time | IQOS Users: 9 Months IQOS Use Time | IQOS Users 12 Months IQOS Use Time | IQOS Users 15 Months IQOS Use Time
Started | 215 | 70 | 191 | 0 | 0 | 0
Completed | 107 | 50 | 191 | 0 | 0 | 0
Not Completed | 108 | 20 | 0 | 0 | 0 | 0
Period: At Month 9
Arm/Group | CC Smokers | IQOS Users: 3 Months IQOS Use Time | IQOS Users: 6 Months IQOS Use Time | IQOS Users: 9 Months IQOS Use Time | IQOS Users 12 Months IQOS Use Time | IQOS Users 15 Months IQOS Use Time
Started | 107 | 50 | 191 | 264 | 0 | 0
Completed | 12 | 42 | 113 | 264 | 0 | 0
Not Completed | 95 | 8 | 78 | 0 | 0 | 0
Period: At Month 12
Arm/Group | CC Smokers | IQOS Users: 3 Months IQOS Use Time | IQOS Users: 6 Months IQOS Use Time | IQOS Users: 9 Months IQOS Use Time | IQOS Users 12 Months IQOS Use Time | IQOS Users 15 Months IQOS Use Time
Started | 12 | 42 | 113 | 264 | 73 | 0
Completed | 4 | 28 | 75 | 134 | 73 | 0
Not Completed | 8 | 14 | 38 | 130 | 0 | 0
Period: At Month 15
Arm/Group | CC Smokers | IQOS Users: 3 Months IQOS Use Time | IQOS Users: 6 Months IQOS Use Time | IQOS Users: 9 Months IQOS Use Time | IQOS Users 12 Months IQOS Use Time | IQOS Users 15 Months IQOS Use Time
Started | 4 | 28 | 75 | 134 | 73 | 1
Completed | 1 | 18 | 31 | 98 | 10 | 1
Not Completed | 3 | 10 | 44 | 36 | 63 | 0
Period: At Month 18
Arm/Group | CC Smokers | IQOS Users: 3 Months IQOS Use Time | IQOS Users: 6 Months IQOS Use Time | IQOS Users: 9 Months IQOS Use Time | IQOS Users 12 Months IQOS Use Time | IQOS Users 15 Months IQOS Use Time
Started | 1 | 18 | 31 | 98 | 10 | 1
Completed | 0 | 6 | 22 | 48 | 7 | 0
Not Completed | 1 | 12 | 9 | 50 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Adult Japanese CC smokers or IQOS users
Groups:
- IQOS Users: The criteria defining a "IQOS user" are listed in the section "Eligibility".
- Total: Total of all reporting groups
Arm/Group | CC Smokers | IQOS Users | Total
Number analyzed (Participants) | 525 | 599 | 1124
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (9.16) | 42.4 (8.67) | 45.0 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 88 | 217
  Male | 396 | 511 | 907
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 525 | 599 | 1124
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 525 | 599 | 1124

OUTCOME MEASURES:

1. Primary Outcome: Product Consumption
Description: To measure the mean numbers of cigarettes smoked and IQOS with HeatSticks used, mean numbers/times of Other Tobacco and Nicotine containing Products (OTP) used. OTP: included all other tobacco and nicotine-containing products except IQOS.
Time Frame: CC smokers: enrollment, IQOS users: 3-18 Months IQOS use time
Population: CC smokers: at enrollment, IQOS users: 3-18 months IQOS use time
Measure: Mean (Standard Deviation); unit: number of consumption per day
Groups:
- IQOS Users: 3 Months IQOS Use; IQOS Users: 6 Months IQOS Use; IQOS Users: 9 Months IQOS Use; IQOS Users: 12 Months IQOS Use; IQOS Users: 15 Months IQOS Use; IQOS Users: 18 Months IQOS Use: The criteria defining a "IQOS user" are listed in the section "Eligibility".
Arm/Group | IQOS Users: 3 Months IQOS Use | IQOS Users: 6 Months IQOS Use | IQOS Users: 9 Months IQOS Use | IQOS Users: 12 Months IQOS Use | IQOS Users: 15 Months IQOS Use | IQOS Users: 18 Months IQOS Use | CC Smokers
Number analyzed (Participants) | 66 | 214 | 375 | 289 | 161 | 84 | 460
number of consumption per day
  Mean number of cigarettes smoked per day | 4.0 (7.72) | 3.8 (6.68) | 4.6 (7.99) | 4.4 (8.12) | 5.1 (8.80) | 4.0 (8.06) | 15.8 (9.43)
  Mean number of Heatsticks used per day | 13.3 (8.85) | 13.2 (7.75) | 13.3 (8.52) | 13.8 (8.68) | 12.7 (8.61) | 12.6 (8.69) | 0.2 (1.93)
  Mean number/times of OTP used per day | 1.8 (6.00) | 2.0 (5.41) | 2.6 (7.97) | 2.5 (7.41) | 2.3 (6.33) | 2.5 (5.84) | 0.5 (2.18)

2. Primary Outcome: Product Use Patterns
Description: To describe product use patterns in CC smokers and IQOS users by product use categories.
  Primarily IQOS: ≥70% consumption of IQOS, Primarily CC: ≥70% consumption of CC, Mixed IQOS-CC: consumption of IQOS in (30% to 70%) AND consumption of CC in (30% to 70%), Mixed IQOS-OTP: consumption of IQOS in (30% to 70%) AND consumption of OTP in (30% to 70%), Mixed CC-OTP: consumption of CC in (30% to 70%) AND consumption of OTP in (30% to 70%), Non-User/smoker: Total consumption of all products = 0, Other: Does not fit in any of the above categories and no 'missing'.
Time Frame: IQOS users: 3-18 months IQOS use, CC smokers from enrollment up to 15 months of follow-up
Population: IQOS users: 3-18 months IQOS use, CC smokers from enrollment up to 15 months of follow-up
Measure: Count of Participants; unit: Participants
Groups:
- CC Smokers Enrollment; CC Smokers After 3 Months Follow-up; CC Smokers After 6 Months Follow-up; CC Smokers After 9 Months Follow-up; CC Smokers After 12 Months Follow-up; CC Smokers After 15 Months Follow-up: The criteria defining a "CC smoker" are listed in the section "Eligibility".
Arm/Group | IQOS Users: 3 Months IQOS Use | IQOS Users: 6 Months IQOS Use | IQOS Users: 9 Months IQOS Use | IQOS Users: 12 Months IQOS Use | IQOS Users: 15 Months IQOS Use | IQOS Users: 18 Months IQOS Use | CC Smokers Enrollment | CC Smokers After 3 Months Follow-up | CC Smokers After 6 Months Follow-up | CC Smokers After 9 Months Follow-up | CC Smokers After 12 Months Follow-up | CC Smokers After 15 Months Follow-up
Number analyzed (Participants) | 70 | 241 | 419 | 310 | 158 | 84 | 525 | 215 | 107 | 12 | 4 | 1
Participants
  Primarily IQOS (≥70% consumption of IQOS) | 45 | 133 | 228 | 182 | 94 | 47 | 2 | 8 | 6 | 2 | 1 | 0
  Primarily CC (≥70% consumption of CC ) | 8 | 16 | 44 | 36 | 26 | 15 | 430 | 204 | 91 | 10 | 3 | 1
  Mixed IQOS-CC (IQOS and CC use in 30% to 70%) | 6 | 29 | 46 | 30 | 15 | 4 | 2 | 2 | 0 | 0 | 0 | 0
  Mixed IQOS-OTP (IQOS and OTP use in 30% to 70%) | 1 | 15 | 22 | 13 | 11 | 12 | 0 | 1 | 1 | 0 | 0 | 0
  Mixed CC-OTP (CC and OTP use in 30% to 70%) | 2 | 4 | 8 | 4 | 3 | 1 | 16 | 7 | 3 | 0 | 0 | 0
  Non-user/Smoker | 0 | 3 | 1 | 1 | 2 | 2 | 7 | 3 | 5 | 0 | 0 | 0
  Other | 4 | 14 | 26 | 23 | 10 | 3 | 3 | 3 | 1 | 0 | 0 | 0
  missing | 4 | 28 | 47 | 23 | 0 | 0 | 65 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Rate of Product Use
Description: To measure the percentage of product use in IQOS users based on IQOS use time.
  * IQOSi = percentage of IQOS use at time point i,
  * CCi = percentage of CC use at time point i,
  * OTPi = percentage of other tobacco products (OTP) use at time point i.
Time Frame: IQOS users: 3-18 months IQOS use time
Population: IQOS users: 3-18 months IQOS use time
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | IQOS Users: 3 Months IQOS Use | IQOS Users: 6 Months IQOS Use | IQOS Users: 9 Months IQOS Use | IQOS Users: 12 Months IQOS Use | IQOS Users: 15 Months IQOS Use | IQOS Users: 18 Months IQOS Use
Number analyzed (Participants) | 70 | 241 | 419 | 310 | 158 | 84
percentage
  % CC | 17.5 (29.0) | 17.0 (27.54) | 19.6 (31.18) | 18.2 (30.34) | 21.7 (34.23) | 19.2 (33.51)
  %OTP | 7.2 (21.42) | 9.3 (22.84) | 9.5 (23.33) | 9.8 (24.89) | 2.3 (6.33) | 2.5 (5.84)
  %IQOS | 75.3 (35.53) | 73.7 (33.62) | 70.9 (36.53) | 72.0 (36.83) | 68.5 (38.81) | 68.9 (37.80)

4. Primary Outcome: Tobacco and Nicotine-containing Products Cessation
Description: To measure rate of cessation from all tobacco and nicotine-containing products in CC smokers and IQOS users
Time Frame: IQOS users: 3-18 months IQOS use time, CC smokers from enrollment up to 15 months of follow-up
Population: IQOS users: 3-18 months IQOS use time, CC smokers from enrollment up to 15 months of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | IQOS Users | CC Smokers
Number analyzed (Participants) | 599 | 525
Participants | 5 | 15

5. Primary Outcome: Demographics of Tobacco and Nicotine-containing Product Users
Description: To describe the demographics characteristics of IQOS users by product use category:
  Primarily IQOS: ≥70% consumption of IQOS, Primarily CC: ≥70% consumption of CC, Mixed IQOS-CC: consumption of IQOS in (30% to 70%) AND consumption of CC in (30% to 70%), Mixed IQOS-OTP: consumption of IQOS in (30% to 70%) AND consumption of OTP in (30% to 70%), Mixed CC-OTP: consumption of CC in (30% to 70%) AND consumption of OTP in (30% to 70%), Non-Use: Total consumption of all products= 0, Other: Does not fit in any of the above categories and no 'missing'.
Time Frame: IQOS users at enrollment
Population: IQOS users at enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Primarily IQOS: ≥70% consumption of IQOS
- Primarily CC: ≥70% consumption of CC
- Mixed IQOS-CC: Consumption of IQOS in (30% to 70%) AND consumption of CC in (30% to 70%)
- Mixed IQOS-OTP: Consumption of IQOS in (30% to 70%) AND consumption of OTP in (30% to 70%)
- Mixed CC-OTP: Consumption of CC in (30% to 70%) AND consumption of OTP in (30% to 70%)
- Non-use: Total consumption of all products=0
- Other: Does not fit in any of the categories and no 'missing'
Arm/Group | Primarily IQOS | Primarily CC | Mixed IQOS-CC | Mixed IQOS-OTP | Mixed CC-OTP | Non-use | Other
Number analyzed (Participants) | 305 | 52 | 64 | 25 | 12 | 1 | 39
Participants
  Male | 263 | 44 | 57 | 22 | 10 | 1 | 37
  20-29 years of age | 20 | 4 | 3 | 1 | 1 | 0 | 4
  30-39 years of age | 102 | 18 | 21 | 9 | 1 | 0 | 11
  40-49 years of age | 128 | 18 | 25 | 11 | 7 | 0 | 11
  50-59 years of age | 50 | 11 | 15 | 2 | 3 | 1 | 12
  60-69 years of age | 4 | 1 | 0 | 2 | 0 | 0 | 0
  70-79 years of age | 1 | 0 | 0 | 0 | 0 | 0 | 1

6. Primary Outcome: Smoking History (Duration)
Description: To record the smoking history (duration) in CC smokers and IQOS users, measured in years.
Time Frame: At enrollment
Population: CC smokers and IQOS users at enrollment
Measure: Mean (Standard Deviation); unit: years
Arm/Group | IQOS Users | CC Smokers
Number analyzed (Participants) | 512 | 492
years | 15.2 (11.84) | 12.0 (13.65)

7. Primary Outcome: Smoking History (Intensity)
Description: To record the smoking history (intensity) in CC smokers and IQOS users, measured in pack-years. One pack year is equivalent to smoking 20 cigarettes a day for one year.
Time Frame: At enrollment
Population: CC smokers and IQOS users at enrollment
Measure: Mean (Standard Deviation); unit: pack years
Arm/Group | IQOS Users | CC Smokers
Number analyzed (Participants) | 524 | 496
pack years | 17.4 (9.12) | 17.0 (10.00)

8. Primary Outcome: Product Usage and Behaviors (Prior to IQOS Use): Smoking Duration
Description: To measure smoking duration among CC smokers who started to use IQOS during follow-up, measured in years.
Time Frame: From enrollment up to 15 months follow-up
Population: CC smokers who started to use IQOS during follow-up
Measure: Mean (Standard Deviation); unit: years
Groups:
- CC Smokers: Subjects enrolled as CC smokers who started to use IQOS during follow-up
Arm/Group | CC Smokers
Number analyzed (Participants) | 21
years | 9.8 (11.47)

9. Primary Outcome: Product Usage and Behaviors (Prior to IQOS Use): Smoking Intensity
Description: To measure smoking intensity among CC smokers who started to use IQOS during follow-up, measured in pack years. One pack year is equivalent to smoking 20 cigarettes a day for one year.
Time Frame: From enrollment up to 15 months follow-up
Population: CC smokers who started to use IQOS during follow-up
Measure: Mean (Standard Deviation); unit: pack years
Arm/Group | CC Smokers
Number analyzed (Participants) | 21
pack years | 13.4 (7.14)

ADVERSE EVENTS:
Time Frame: 15 Months
Description: As this study was observational by design and was conducted in a post-market setting, adverse event (AE) reporting followed the Sponsor's established post-market Safety Surveillance Procedures for spontaneously reported events. IQOS users were reminded of the product quality complaints (including AEs) hotline that is available for all IQOS consumers in Japan.
Groups:
- All Participants: All subjects that participated in the study.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/1124
Serious Adverse Events (participants affected / at risk) | 0/1124
Other Adverse Events (participants affected / at risk) | 0/1124

LIMITATIONS AND CAVEATS:
Due to study termination leading to a shortened follow-up period and a smaller sample size, only 7 outcome measures could be assessed and the other outcome measures originally planned were either unattainable or uninformative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT03020667/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT03020667/SAP_001.pdf